CLINICAL TRIAL: NCT01335373
Title: Observational Program Neo-Penotran® Forte
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15511; NP1010KZ (Other: company internal)
Record Dates: First submitted 2011-01-21; First posted 2011-04-14 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-05

CONDITIONS: Vaginal Candidiasis; Bacterial Vaginosis; Trichomonal Vaginitis
Keywords: Vaginal candidiasis; Bacterial vaginosis (also known as non-specific, or Gardnerellosis, or anaerobic vaginosis); Trichomonal vaginitis; Vaginitis due to mixed infection
MeSH Terms: conditions — Candidiasis, Vulvovaginal; Vaginosis, Bacterial; Trichomonas Vaginitis | interventions — Metronidazole; Miconazole

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Metronidazole/Miconazole (Neo-Penotran Forte, BAY86-5276)

INTERVENTIONS:
Drug: Metronidazole/Miconazole (Neo-Penotran Forte, BAY86-5276) — Patients older than 18 years with previously taken decision of their gynecologist to prescribe Neo-Penotran Forte according to registered indications, and microbiological tests were performed.

SUMMARY:
Vaginitis is the most common gynecologic diagnosis in the primary care setting. In approximately 90 percent of affected women, this condition occurs secondary to bacterial vaginosis, vulvovaginal candidiasis, trichomoniasis or mixed infection.

Neo-Penotran Forte is registered for treatment of these most common vaginal infections. Efficacy and safety of this product is already established, and this observational study was designed to learn more about practical use of Neo-Penotran® Forte in real life setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years with previously taken decision of their gynecologist to prescribe Neo-Penotran Forte according to registered indications, and microbiological tests were performed.

Exclusion Criteria:

* Presence of contraindications according to package insert.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in primary care setting.
Sampling Method: Non-Probability Sample
Enrollment: 13024 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percent rate of different vaginal infections | Approximately within 6 months after the last patient last visit.

SECONDARY OUTCOMES:
Clinical characteristics of vaginitis after treatment. | Depending on treatment time chosen by the physician, after 7 or 14 days.
Change of microbiological characteristics after treatment | Depending on treatment time chosen by the physician, after 7 or 14 days.
Patient rating of tolerability and treatment results | Depending on treatment time chosen by the physician, after 7 or 14 days.
Physician's rating of tolerability and treatment results | Depending on treatment time chosen by the physician, after 7 or 14 days.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Kazakhstan